CLINICAL TRIAL: NCT04241094
Title: Teaching Loved Ones to Help Veterans Optimize Their PTSD Care and Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3460-P
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Couples therapy; Psychotherapy; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Loved one assisted treatment (Experimental): The investigators propose to bring a loved one into PE, one of the most researched and efficacious treatments for PTSD, to increase support for PE adherence. The intervention is a 13-session cognitive-behavioral, intimate partner-assisted treatment for PTSD that draws from PE, ICBT, and PE2.
  Interventions: Behavioral: Loved one assisted treatment

INTERVENTIONS:
Behavioral: Loved one assisted treatment — The investigators propose to bring a loved one into PE, one of the most researched and efficacious treatments for PTSD, to increase support for PE adherence. The intervention is a 13-session cognitive-behavioral, intimate partner-assisted treatment for PTSD that draws from PE, ICBT, and PE2.

SUMMARY:
PTSD occurs in as many as 17% of US military Veterans and is associated with a host of negative, long-term consequences to the individual, their families, and society at large. EBPs, such as Prolonged Exposure, result in clinically significant symptom relief for many. Yet, these therapies have proven less effective for military personnel and Veterans and treatment dropout rates are high. The investigators' team surveyed Veterans initiating EBPs for PTSD and a family member across four VA medical centers (N = 598; Project HomeFront). The investigators found that Veterans were more than twice as likely to complete EBPs when loved ones encouraged them to confront distress and that Veterans experienced greater treatment gains when they shared more with their loved ones about their treatment. A couples-based, exposure therapy for PTSD that integrates intimate partners into every session of PE could provide the opportunity to mobilize the whole household in the service of EBP engagement, while extending the goals of therapy beyond symptom reduction to family functioning. The investigators anticipate this intervention will teach couples to embrace a lifestyle that supports confronting trauma-related distress, so the Veteran and his/her family can achieve optimal functional outcomes.

DETAILED DESCRIPTION:
The investigators aim to improve the mental health, family functioning, and well-being of Veterans with posttraumatic stress disorder (PTSD) through developing and evaluating a trauma-focused, couple therapy for PTSD. The investigators will use strategies from Integrative Behavioral Couple Therapy (ICBT) to help intimate partners support Veterans during exposure therapy for PTSD (Prolonged Exposure; PE). The investigators anticipate this approach will increase Veterans' engagement in PE, but also improve relationship functioning, family functioning, and social functioning. Family involvement has been highlighted as a fertile avenue for improving the outcomes for patients with PTSD, yet families are infrequently integrated into evidence-based psychotherapies (EBPs). The investigators' goals are highly consistent with RR&D's mission to promote research that leverages family support as a pathway to reintegration and optimizes meaningful recovery and functioning.

Objectives. The investigators will complete stages 1A and 1B of the Stage Model of Treatment Development. Specifically, the investigators will: (1) Expand the treatment outline using content experts and feedback from key stakeholders (Veterans, intimate partners, providers, and VA mental health leadership). (2) Conduct a pilot open trial to assess (a) the acceptability of treatment components, structure, and materials, (b) the feasibility of the intervention (retention and intervention fidelity), and (c) the study approach (screening, recruitment, and assessment process). (3) Explore the preliminary effects of the intervention on select outcomes including overall functioning, mental health functioning, social functioning, family functioning, and potential mechanisms (social control, subjective norms, and the degree to which Veterans rely on their partners for support).

Methods: To accomplish Aim 1, the investigators will expand the outline for the intervention into an initial treatment manual through meetings with content experts and stakeholder feedback. Next, the investigators will develop fidelity checklists and revise the treatment manual through conducting the intervention with 2-3 couples. To accomplish Aims 2 and 3, the investigators will evaluate the intervention in a non-randomized, open trial with 10 Veterans diagnosed with PTSD and their intimate partners. Veterans will complete baseline and posttreatment structured diagnostic interviews. Both members of the couple will complete baseline surveys, posttreatment surveys, and posttreatment qualitative exit interviews. Using data obtained from the open trial, the investigators will assess the intervention's acceptability, feasibility, mechanisms, and outcomes. Upon completion of this proposal, the investigators will be well positioned to apply for Merit funding for a randomized clinical trial (Stage 2 of the Stage Model of Treatment Development) of this innovative, exposure based, couple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in VHA care
* Clinically significant PTSD symptoms
* Have a LO (loved one/intimate partner) with whom they have been in a romantic relationship with for 6 months
* Will allow a LO to participate
* Willing to be seen via telehealth when in-person treatment options aren't available.

Exclusion Criteria:

* Actively suicidal/homicidal with intent and/or plan
* Episode of mania/ psychosis in past 3 months
* Severe substance use problem in past 3 months
* Moderate relationship violence
* Veteran has underlying medical condition or a planned medical procedure likely to impair ability to engage in treatment.
* LO screens positive for PTSD
* Veteran and/or LO fails to complete baseline survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Meis, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (3):
- United States (3):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 Veterans were consented and signed informed consent for the study. Only 20 of those 28 went forward with the COACH treatment.
Pre-assignment Details: The numbers in this chart are counted as individual participants. 28 participants (16 Veterans and 12 loved ones) consented to the study. Of those 28, only 20 participants (10 Veterans and 10 loved ones) started treatment in the study.
Period: Overall Study
Arm/Group | Loved One Assisted Treatment
Started | 20 (Started treatment)
Never Started Treatment (These Veteran were enrolled, but never began the COACH treatment) | 8
Completed | 12 (Completed treatment)
Not Completed | 8
Not completed — Dropped out of treatment | 4
Not completed — Ineligible after clinical assessment | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The numbers in this chart are counted as individual participants. 28 participants (16 Veterans and 12 loved ones) consented to the study. Of those 28, only 20 participants (10 Veterans and 10 loved ones) started treatment in the study. Baseline data characteristics were collected for both Veterans and loved ones.
Arm/Group | Loved One Assisted Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants] — Population: There are two cohort types in this study: Veterans and loved ones
  Participants
    Veterans: number analyzed (Participants) | 10
    Veterans: <=18 years | 0
    Veterans: Between 18 and 65 years | 10
    Veterans: >=65 years | 0
    Loved Ones: number analyzed (Participants) | 10
    Loved Ones: <=18 years | 0
    Loved Ones: Between 18 and 65 years | 10
    Loved Ones: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are two cohort types in this study: Veterans and loved ones
  Participants
    Veterans: number analyzed (Participants) | 10
    Veterans: Female | 4
    Veterans: Male | 6
    Loved ones: number analyzed (Participants) | 10
    Loved ones: Female | 7
    Loved ones: Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: There are two cohort types in this study: Veterans and loved ones
  Participants
    Veterans: number analyzed (Participants) | 10
    Veterans: Hispanic or Latino | 0
    Veterans: Not Hispanic or Latino | 10
    Veterans: Unknown or Not Reported | 0
    Loved ones: number analyzed (Participants) | 10
    Loved ones: Hispanic or Latino | 0
    Loved ones: Not Hispanic or Latino | 10
    Loved ones: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There are two cohort types in this study: Veterans and loved ones
  Participants
    Veterans: number analyzed (Participants) | 10
    Veterans: American Indian or Alaska Native | 1
    Veterans: Asian | 0
    Veterans: Native Hawaiian or Other Pacific Islander | 0
    Veterans: Black or African American | 0
    Veterans: White | 8
    Veterans: More than one race | 1
    Veterans: Unknown or Not Reported | 0
    Loved ones: number analyzed (Participants) | 10
    Loved ones: American Indian or Alaska Native | 0
    Loved ones: Asian | 1
    Loved ones: Native Hawaiian or Other Pacific Islander | 0
    Loved ones: Black or African American | 0
    Loved ones: White | 8
    Loved ones: More than one race | 1
    Loved ones: Unknown or Not Reported | 0
Length of relationship [Count of Participants; unit: Participants] — Population: There are two cohort types in this study: Veterans and loved ones
  Participants
    Veterans: number analyzed (Participants) | 10
    Veterans: 6+ months | 1
    Veterans: 1-4 years | 3
    Veterans: 5-10 years | 3
    Veterans: 11+ years | 3
    Loved ones: number analyzed (Participants) | 10
    Loved ones: 6+ months | 1
    Loved ones: 1-4 years | 3
    Loved ones: 5-10 years | 3
    Loved ones: 11+ years | 3

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale for DSM-5 to Assess Changes in PTSD Symptoms.
Description: Structured clinical interview assessing symptoms of PTSD. CAPS-5 is a 30-item questionnaire, corresponding to the DSM-5 diagnosis for PTSD. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. Similarly, CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. Severity scores range from 0 to 80 and higher scores correspond with more severe symptoms of PTSD.
Time Frame: Up to 26 weeks post baseline
Population: Veteran participants
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Loved One Assisted Treatment at Baseline: The investigators propose to bring a loved one into PE, one of the most researched and efficacious treatments for PTSD, to increase support for PE adherence. The intervention is a 13-session cognitive-behavioral, intimate partner-assisted treatment for PTSD that draws from PE, ICBT, and PE2.
  Loved one assisted treatment: The investigators propose to bring a loved one into PE, one of the most researched and efficacious treatments for PTSD, to increase support for PE adherence. The intervention is a 13-session cognitive-behavioral, intimate partner-assisted treatment for PTSD that draws from PE, ICBT, and PE2. This is data from Veterans before treatment begins.
- Loved One Assisted Treatment at Posttreatment: The investigators propose to bring a loved one into PE, one of the most researched and efficacious treatments for PTSD, to increase support for PE adherence. The intervention is a 13-session cognitive-behavioral, intimate partner-assisted treatment for PTSD that draws from PE, ICBT, and PE2.
  Loved one assisted treatment: The investigators propose to bring a loved one into PE, one of the most researched and efficacious treatments for PTSD, to increase support for PE adherence. The intervention is a 13-session cognitive-behavioral, intimate partner-assisted treatment for PTSD that draws from PE, ICBT, and PE2. This is data from Veterans after treatment ended.
Arm/Group | Loved One Assisted Treatment at Baseline | Loved One Assisted Treatment at Posttreatment
Number analyzed (Participants) | 10 | 6
score on scale | 35.3 (9.12) | 11.33 (7.26)

ADVERSE EVENTS:
Time Frame: The investigators collected adverse event data for all participants (Veterans and loved ones) from the date of enrollment through date of 3 month follow-up assessment. This included reviewing the medical chart for all veteran participants. For loved ones, the investigators would include adverse events that were explicitly stated by loved ones to study staff (none of these occurred).
Description: This is a minimal risk study with very few participants. The likelihood of a serious adverse event or death is not likely.
Arm/Group | Loved One Assisted Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04241094/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04241094/ICF_000.pdf